CLINICAL TRIAL: NCT04939194
Title: Fast Track Protocol After Radical Cystectomy and Urinary Diversion: A Randomised Controlled Trial.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Lashin, A.M.Lashin, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNC , Mansoura
Record Dates: First submitted 2021-06-16; First posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Bladder Cancer
Keywords: ERAS (Early Recovery After Surgery); Radical Cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast Track Protocol (Experimental): the 22 items of ERAS (Early Recovery After Surgery) society
  Interventions: Behavioral: Fast Track Protocol
- Conventional perioperative care program (No Intervention): standard perioperative care

INTERVENTIONS:
Behavioral: Fast Track Protocol — We will apply 22 items of ERAS society
  Arms: Fast Track Protocol

SUMMARY:
We will design a randomized controlled single center study in which we will compare 2 groups of patients, 1 with standard perioperative protocols and another one in which we will apply fast track protocols in patients after radical cystectomy and urinary diversion .

DETAILED DESCRIPTION:
Study hypothesis:

Fast Track Protocol after Radical Cystectomy reduces the length of hospital stay and the early postoperative complications relative to the traditional perioperative care regimen.

Purpose of the study:

1. To evaluate the the perioperative efficacy, safety and benefits of fast track protocol implementation after radical cystectomy and to optimize perioperative patient care for the benefit of "fast-track" surgery.
2. To evaluate early complications in patients with bladder cancer who will be subjected to radical cystectomy and urinary diversion.

Study groups:

Group 1: Fast Track group (105 patients). Group 2: Conventional perioperative care group (105 patients).

Study design:

The design of the research will be a prospective randomised, open-label, controlled study on 210 consecutive patients with bladder cancer who will be subjected to radical cystectomy and urinary diversion. All the patients will sign an informed consent. Length of stay, dietary issues, and return of bowel function, readmission rates and complications will be evaluated.

Study setting/location:

The study will be conducted in a single tertiary centre, Urology and Nephrology Centre in Mansoura, Egypt. The study will be carried out on patient with bladder cancer who will be subjected to radical cystectomy and urinary diversion.

Study duration:

The study will last about 2 and half years.

Randomisation:

Randomization will be performed using computer generated, sequentially numbered random tables. Ratio of assignment to groups is 1: 1.

Allocation concealment and blinding:

We are well aware that it is very difficult to properly blind trials comparing surgical treatments. Allocation of patients to treatment groups will be self-evident following randomization and blinding of patient groups and observers will not be possible. So, our trial will be a randomised, open-label, controlled trial.

Type of analysis:

Intention-to-treat analysis is planned in this trial. We will include all patients randomized to the fast track group regardless of their adherence and compliance to the early recovery after surgery (ERAS) items.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing radical cystectomy and urinary diversion surgery including orthotopic neobladder and ileal loop conduit

Exclusion Criteria:

1. Radical cystectomy performed in an emergency setting
2. Patients who refused fast track protocol
3. Mental illnesses

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay. | 3 months after surgery.
  Mean length of hospital stay defined as days from admission to the hospital, in both groups 1 day before surgery and discharge.

SECONDARY OUTCOMES:
Early postoperative complications rate defined and graded according to Clavien-Dindo system. | 3 months after surgery.
  Rate of early postoperative complications eg: anastomotic leakage, intestinal obstruction, wound infection.
Hospital readmission rate. | 3 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mosbah, Prof., Study Chair — Urology department , Urology and Nephrology Center , Faculty of Medicine, Mansoura University, Egypt; Mahmoud Laymon, Lecturer., Study Director — Urology department , Urology and Nephrology Center , Faculty of Medicine, Mansoura University, Egypt; Ahmed Lashin, Dr., Principal Investigator — Urology department , Urology and Nephrology Center , Faculty of Medicine, Mansoura University, Egypt
Locations (1):
- Mansoura Urology & Nephrology Center, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No